CLINICAL TRIAL: NCT05248490
Title: Impact of Pharmaceutical Interviews Regarding the Management of Adverse Effects Related to the Antibiotic Therapy Used to Treat Osteoarticular Infections During Return Home
Acronym: EFIRAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP211422; 2021-A02433-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-01-21; First posted 2022-02-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Bone and Joint Infection
Keywords: osteo articular infection; adverse event; antibiotic treatment; pharmaceutical interview

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with pharmaceutical interview (Experimental): Pharmaceutical interview with pharmacist: to be informed treatment taken and related SAE informations at the end of hospitalization.
  Interventions: Other: pharmaceutical interview
- Patients without pharmaceutical interview (No Intervention): Control group without interview

INTERVENTIONS:
Other: pharmaceutical interview — Pharmaceutical interview with pharmacist: to be informed treatment taken and related SAE informations at the end of hospitalization
  Arms: Patients with pharmaceutical interview

SUMMARY:
The primary objective is to evaluate the impact of Pharmaceutical Interviews in the patient self-management of non-severe side effects caused by antibiotics prescribed for the treatment of osteoarticular infections when the patient returns home.

ELIGIBILITY:
Inclusion Criteria:

* Patient > or =18 years;
* Informed consent signed;
* French-speaking and reading;
* Affiliated to a social insurance;
* Benefiting from medical and surgical care for an osteoarticular infection;
* Treated with an oral antibiotic therapy on discharge from hospital.
* Indication of the antibiotic therapy osteoarticular infection;
* Return home immediately after discharge.

Exclusion Criteria:

* Refusal to participate
* Protected adult patient, under guardianship or curatorship.
* Minor patient
* Patient benefiting from an AME.
* Pregnant or breastfeeding woman.
* Non-French speaking patient.
* Patient unable to understand the course of the study.
* Patient with a documented history of cognitive or psychiatric disorders.
* Patient treated with oral antibiotic therapy for an indication other than osteoarticular infection.
* Patient treated with parenteral antibiotic therapy.
* Discharge: Institution (EHPAD), rehabilitation or other health establishment.
* Patient systematically using one of the symptomatic treatments proposed in the discharge prescription before hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Adverse effects self-management measurement | at day 7
  Phone call to evaluate the self-management of adverse effects. Self-management evaluation (optimal choice/non-optimal choice) performs thanks to the use of a standardized decision-tree.
  Proportion of patients with an optimal or non-optimal self-management.
Adverse effects self-management measurement | at day 14
  Phone call to evaluate the self-management of adverse effects. Self-management evaluation (optimal choice/non-optimal choice) performs thanks to the use of a standardized decision-tree.
  Proportion of patients with an optimal or non-optimal self-management.

SECONDARY OUTCOMES:
Patient knowledge assessment | at day 7
  Questionnaire, 12 points:
  * proportion of patients reaching a score upper than 10
  * proportion of patients reaching a score between 6 and 9
  * proportion of patients reaching a score lower than 6

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tritz, PharmD, Principal Investigator — Pharmacy of Ambroise-Paré hospital, APHP; Christophe Menigaux, MD, Study Chair — Orthopedic surgery department, Ambroise Paré hospital, APHP; Nathalie Dournon, MD, Study Chair — Infectiology mobile team, Ambroise Paré hospital, APHP; Jessica Berdougo Berdougo, PharmD, Study Chair — Pitié-Salepetrière hospital, APHP
Locations (1):
- Pharmacy of Ambroise-Paré hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No